CLINICAL TRIAL: NCT03025932
Title: Clinical vs. Radiological Recurrence Rate After Laparoscopic Repair of Large Hiatal Hernia With Mesh and Anterior Fundoplication
Brief Title: Recurrence Rate After Laparoscopic Repair of Large Hiatal Hernia
Status: Enrolling by invitation | Type: Observational
Sponsor: Prof Urs Zingg (Other)
Responsible Party: Sponsor-Investigator, Prof Urs Zingg, PD Dr. med., Spital Limmattal Schlieren
Organization: Spital Limmattal Schlieren (Other)
Other Study IDs: 2016-01510
Record Dates: First submitted 2017-01-09; First posted 2017-01-20 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Hiatal Hernia Large
MeSH Terms: interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient cohort: Patients who underwent laparoscopic hernia repair of giant hiatal hernia with mesh and received anterior fundoplication
  Interventions: Procedure: repair of giant hiatal hernia with mesh and anterior fundoplication

INTERVENTIONS:
Procedure: repair of giant hiatal hernia with mesh and anterior fundoplication

SUMMARY:
Patients who underwent laparoscopic repair of large hiatal hernias and anterior fundoplication with mesh are examined for their recurrence rate one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Initially suffering from large hiatal hernia (>20% of the stomach in the thoracic cavity)
* Performance of laparoscopic hiatal hernia repair with mesh and anterior fundoplication
* Informed Consent as documented by signature (Appendix: Informed Consent Form)

Exclusion Criteria:

* Performance of any other anti-reflux surgery such as Toupet- or Nissen-fundoplication
* Performance of anterior fundoplication without mesh
* Women who meet the inclusion criteria but are pregnant or breast feeding or have the intention to become pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion of all patients older than 18 years with initial large hiatal hernia (>20% herniated into thoracic cavity) and laparoscopic hiatoplasty with mesh and anterior fundoplication
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Radiological recurrence rate of hiatal hernia determined by computer tomography (CT) scan | minimum 1 year after surgery
  To evaluate the radiological recurrence rate of hiatal hernia at least one year after surgery by performing a computer tomography

SECONDARY OUTCOMES:
Quality of life by GIQLI | minimum 1 year after surgery
  Estimate the quality of life using a standardized questionnaire (Gastrointestinal Qualitiy of Life Index = GIQLI) at least one year after surgery
Clinical outcome | minimum 1 year after surgery
  Evaluate the clinical outcome at least one year after surgery by examining the patient and asking targeted questions on the symptoms regarding the former hiatal hernia (using visual analogue scale questions on dysphagia, meteorism, bloating, reflux and retrosternal pain). Furthermore the patients are asked about their general satisfaction regarding the performed surgical intervention.
Peri- and postoperative morbidity / mortality | minimum 1 year after surgery
  Evaluate the peri- and postoperative morbidity and mortality from the patient records and a clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Urs Zingg, Principal Investigator — Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Susstrunk J, Stimpfle D, Wilhelm A, Ghielmini EM, Potthast S, Zingg U. Clinical and computed tomography outcomes after mesh-enforced hiatoplasty and anterior hemi-fundoplication in large hiatal hernia repair. World J Surg. 2024 Nov;48(11):2669-2677. doi: 10.1002/wjs.12354. Epub 2024 Sep 20. PMID 39304965